CLINICAL TRIAL: NCT03183453
Title: Replica Study of a Neuropsychological Treatment for Patients Who Show Spontaneous Confabulation After Acquired Brain Injury
Brief Title: Neuropsychological Rehabilitation of Spontaneous Confabulation: a Replica Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monica Triviño Mosquera (Other)
Responsible Party: Sponsor-Investigator, Monica Triviño Mosquera, Psychology PhD, San Rafael University Hospital, Granada, Spain
Organization: San Rafael University Hospital, Granada, Spain (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Conf-02
Record Dates: First submitted 2017-04-25; First posted 2017-06-12 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Memory Disorders
Keywords: Confabulations; Neuropsychological rehabilitation; Memory
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neuropsychological treatment (Experimental): The tested treatment is a combination of neuropsychological rehabilitation procedures: learning, episodic memory recall after a delay, selective attention, inhibition of predominant responses and awareness of deficits.
  Interventions: Behavioral: Neuropsychological treatment
- Non-confabulators control group (No Intervention): Non-confabulators (brain injured patients but without confabulations) in this control group only performed the pre- and post-measurements without treatment.
- Healthy control group (No Intervention): Healthy participants in this control group only performed the pre- and post-measurements without treatment.

INTERVENTIONS:
Behavioral: Neuropsychological treatment — Participants had to learn some brief material (words, faces, pictures, news), after which they were asked for an immediate and a delayed recall. After both recalls, participants were confronted with feedback about correct responses, non-responses and errors (i.e., confabulations and errors of attribution). This type of feedback worked on: 1) selective attention during the learning phase, training patients to focus on the relevant details of the stimuli; 2) monitoring processes during the retrieval phase, reinforcing the strategic search and training patients to inhibit traces that were irrelevant; and 3) memory control processes after the retrieval phase. The treatment consisted of 9 sessions and lasted for 3 weeks and the participants performed a baseline before and after treatment.
  Other Names: Confabulations treatment
  Arms: Neuropsychological treatment

SUMMARY:
Confabulators consistently generate false memories without intention to deceive and with great feeling of rightness. However, there is currently no known effective treatment for them. In order to fill this gap, we performed a neuropsychological treatment in two groups of confabulators: experimental vs. control (ClinicalTrials.gov ID: NCT02540772).

Now, we intend to replicate the treatment with a larger sample of confabulators and with other two control groups: non-confabulator patients with brain injury and healthy individuals

DETAILED DESCRIPTION:
The treatment consisted of some brief material that patients had to learn and recall at both immediate and delayed moments. After both recollections, patients were given feedback about their performance (errors and correct responses). Pre-treatment and post-treatment measurements were administered.

Non-confabulator patients and healthy participants performed only the pre-treatment measurement.

ELIGIBILITY:
Inclusion Criteria:

* The presence of spontaneous confabulations after acute brain injury, for at least three months and without clinical improvement (interfering with the patient's daily life with frequent arguments and exhaustive supervision).
* The presence of momentary confabulations in the Spanish adaptation of Dalla Barba provoked confabulation interview.
* Prior to injury, all patients should be completely independent for daily living.

Exclusion Criteria:

* The presence of impairment in alertness.
* Dementia.
* Acute confusional state.
* A history of drug abuse.
* Psychiatric antecedents.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change in the number of Confabulations | A first measure (pre-treatment) was recorded after the recruitment up maximum to 1 month. A second measure (post-treatment) after 3 weeks (that was the duration of the treatment).
  The confabulations recorded were 1) guessed answers, 2) confusions in time and space, 3) a mixture of two or more stimuli presented, and 4) devised or bizarre responses.
  Scores ranged from 0 (no confabulations) to unlimited number of them (because devised or bizarre responses were recorded) and consisted of the sum of all the confabulations produced during the 3 sessions.
Change in the number of correct responses | A first measure (pre-treatment) was recorded after the recruitment up maximum to 1 month. A second measure (post-treatment) after 3 weeks (that was the duration of the treatment).
  Scores ranged from 0 (no correct answers) to 72 (12 stimuli remembered twice in each session: firstly, in a immediate recall after learning, and secondly, in a delayed recall after 10 minutes).
Change in the number of non-responses | A first measure (pre-treatment) was recorded after the recruitment up maximum to 1 month. A second measure (post-treatment) after 3 weeks (that was the duration of the treatment).
  Scores ranged from 0 (no non-responses) to 72 (12 stimuli remembered twice in each session: firstly, in a immediate recall after learning, and secondly, in a delayed recall after 10 minutes).

SECONDARY OUTCOMES:
Change in the number of errors in source attribution | A first measure (pre-treatment) was recorded after the recruitment up maximum to 1 month. A second measure (post-treatment) after 3 weeks (that was the duration of the treatment).
  After the recall of the material, patients were also asked to remember which modality corresponded to each recall (i.e., seen, heard or imagined), and who had presented the material during the learning session (i.e., the therapist or themselves).
  Scores ranged from 0 (if all answers were non-responses) to unlimited number (depending on number of confabulations produced by patients).

CONTACTS AND LOCATIONS:
Overall Officials: Monica Triviño, PhD, Principal Investigator — San Rafael University Hospital
Locations (1):
- San Rafael University Hospital, Granada, Spain

REFERENCES:
- [Background] Gilboa A, Alain C, Stuss DT, Melo B, Miller S, Moscovitch M. Mechanisms of spontaneous confabulations: a strategic retrieval account. Brain. 2006 Jun;129(Pt 6):1399-414. doi: 10.1093/brain/awl093. Epub 2006 Apr 25. PMID 16638795
- [Background] Trivino M, Rodenas E, Lupianez J, Arnedo M. Effectiveness of a neuropsychological treatment for confabulations after brain injury: A clinical trial with theoretical implications. PLoS One. 2017 Mar 3;12(3):e0173166. doi: 10.1371/journal.pone.0173166. eCollection 2017. PMID 28257420
- [Background] Schnider A. The confabulating mind. How the brain creates reality. Oxford: Oxford University Press; 2008
- [Background] Nahum L, Bouzerda-Wahlen A, Guggisberg A, Ptak R, Schnider A. Forms of confabulation: dissociations and associations. Neuropsychologia. 2012 Aug;50(10):2524-34. doi: 10.1016/j.neuropsychologia.2012.06.026. Epub 2012 Jul 7. PMID 22781813
- [Background] Ciaramelli E, Ghetti S, Borsotti M. Divided attention during retrieval suppresses false recognition in confabulation. Cortex. 2009 Feb;45(2):141-53. doi: 10.1016/j.cortex.2007.10.006. Epub 2008 Feb 6. PMID 19150516